CLINICAL TRIAL: NCT05498012
Title: Cannabidiol Effects on Chronic Periodontitis: Monocentric, Randomized, Interventional and Placebo-controlled Study
Brief Title: CBD Effects on Periodontal Health of Patients With Chronic Periodontitis
Acronym: Stoma-CBD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Palacky University (Other)
Collaborators: CB21 Pharma Ltd. (Unknown)
Responsible Party: Principal Investigator, Jan Vacek, Department of Dentistry, Olomouc University Hospital, Palacky University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: #3620
Record Dates: First submitted 2022-03-16; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Chronic Periodontitis
Keywords: Periodontitis; Phytocannabinoid; Cannabidiol; Dental gel; Oral microbiota; Inflammation
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): Dental gel applied by dentist after oral hygiene (no cannabidiol). Toothpaste for daily use as needed for patients (no cannabidiol).
  Interventions: Combination Product: placebo dental gel, placebo toothpaste
- CBD group (Experimental): Dental CBD (cannabidiol) gel applied by dentist after oral hygiene. CBD toothpaste for daily use as needed for patients.
  Interventions: Combination Product: Cannabidiol dental gel, Cannabidiol toothpaste
- Corsodyl group (Active Comparator): Corsodyl dental gel applied by dentist after oral hygiene. Toothpaste for daily use as needed for patients (no cannabidiol).
  Interventions: Combination Product: Placebo toothpaste, Corsodyl dental gel

INTERVENTIONS:
Combination Product: placebo dental gel, placebo toothpaste — * Placebo dental gel applied by dentist after oral hygiene; without cannabidiol.
  * Placebo toothpaste; without cannabidiol. For daily use by patient.
  Arms: Placebo group
Combination Product: Cannabidiol dental gel, Cannabidiol toothpaste — * Cannabidiol dental gel applied by dentist after oral hygiene; containing 1 % (w/w) cannabidiol.
  * Cannabidiol toothpaste; containing 1 % (w/w) cannabidiol. For daily use by patient.
  Arms: CBD group
Combination Product: Placebo toothpaste, Corsodyl dental gel — * Corsodyl dental gel; containing 1 % (w/w) chlorhexidini digluconatis applied by dentist after oral hygiene.
  * Placebo toothpaste; without cannabidiol. For daily use by patient.
  Arms: Corsodyl group

SUMMARY:
The suppression of chronic periodontitis after application of dental gel and toothpaste containing cannabidiol (CBD) will be evaluated.

DETAILED DESCRIPTION:
Current state of the art: Non-psychotropic cannabinoids (especially cannabidiol, CBD) are used as drugs and anti-inflammatory components in a number of medical devices. Their use in dentistry (in the form of a full-fledged clinical trial) has not yet been tested. Several pharmacological activities have recently been demonstrated for CBD. Its anti-inflammatory and anti-bacterial action on oral cavity tissues may be beneficial for patients after dental surgery or in patients with periodontal problems. To date, the only registered clinical trial with CBD as the active ingredient in toothpaste and mouthwash was conducted at Swinburne University of Technology in Melbourne (ANZCTR 2019). The products are tested on men aged from 18 to 30 years with chronic gingivitis diagnosis.

Study description: The aim of the study is to evaluate the effect of CBD on the periodontal disease. The study will be conducted as a 67-day, monocentric, randomized, interventional, and placebo-controlled clinical trial. The effect of dental gel and toothpaste containing CBD will be tested. The main evaluated criteria will include a series of periodontal and hygienic indices. The study will be carried out in accordance with the Helsinki Declaration of Human Rights and CONSORT rules.

Recruitment and study design: Recruitment (men and women, age 35-65) will be followed by several visits:

1. At the first visit (0 day), patients who meet the inclusion criteria will be documented via the set of periodontal, gingival and hygienic indices, microbiological sampling, removal of supra/sub-gingival plaque and calculus will be done. Furthermore, a gingival sample will be collected for histopathological examination and, hygienic instructions will take place.
2. At the second visit (day 7), the patients will be checked for proper oral hygiene, patient's periodontal health will be assessed via the set of periodontal, gingival and hygienic indices and CBD dental gel (or identical placebo without CBD) will be applied (5 min exposure). Toothpastes containing CBD or placebo will be handed over. The patients will use the toothpastes to substitute their normal dental hygiene for the duration of the study.
3. At the third visit (day 22), patient's periodontal health will be assessed via the set of periodontal, gingival and hygienic indices and CBD dental gel (or identical placebo without CBD) will be applied (5 min exposure).
4. At the fourth visit (day 37), in case of termination of therapy, gingival samples will be collected for histopathological examination. Patient's periodontal health will be assessed via the set of periodontal, gingival and hygienic indices. A microbiological sample will be collected as well. If the therapy is continued, hygienic re-instruction and repeated application of CBD gel will take place (5 min exposure).
5. During the last visit, patient's periodontal health will be assessed via the set of periodontal, gingival and hygienic indices. Microbiological sampling will be performed. The total duration of the study was set at 67 days.

Evaluation of study results: The clinical study will be evaluated based on measurement of Russell's periodontal index, plaque index and gingival index, gingival bleeding index and modified gingival index. Statistical analysis will be performed in SPSS or STATA software. Furthermore, microbiological sampling and gingival samples for histopathological examination (count of plasmocytes, T-lymphocytes, B-lymphocytes and macrophages in interdental papilla) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Chronic periodontitis
* Age 35-65 years
* Number of native teeth 16 or 16+
* Signed informed consent
* Without physical or mental impairment

Exclusion Criteria:

* Chronic diseases (diabetes mellitus, oncological diseases)
* Increased bleeding (medications - anticoagulants, antiplatelet agents, bleeding diathesis)
* Pregnant and lactating women
* Tabacco smokers
* Users of cannabis or cannabis products
* ATB treatment during the last 3 months
* Patient with removable prosthesis
* Parallel participation in another clinical trial

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Effect of cannabidiol on periodontal health (Russell's periodontal index ) of patients with chronic periodontitis | Baseline (0 day) and 67 days
  Subjects will undergo the measurement of periodontal index according to A.L. Russell.
  Data will be collected based on five possible clinical conditions corresponding to the following scoring:
  Score 0-0.2 (clinical normally supportive tissue) Score 0.3-0.9 (simple gingivitis) Score 1.0-1.9 (beginning destructive periodontal disease) Score 2.0-4.9 (established destructive periodontal disease) Score 5.0-8.0 (terminal disease)
  Change = (Score after 67 days - Baseline score)
Effect of cannabidiol on periodontal health (plaque/gingival indices) of patients with chronic periodontitis | Baseline (0 day) and 67 days
  Subjects will undergo the measurement of plaque/gingival indeces according to H. Löe. Data will be collected based on clinical conditions corresponding to the following scoring systems:
  Plaque index:
  Score 0 (excellent) Score 0.1-0.9 (good) Score 1.0-1.9 (fair) Score 2.0-3.0 (poor)
  Gingival index:
  Score 0.1-1 (mild inflammation) Score 1.1-2 (moderate inflammation) Score 2.1-3 (severe inflammation)
  Change = (Score after 67 days - Baseline score)
Effect of cannabidiol on periodontal health (bleeding) of patients with chronic periodontitis | Baseline (0 day) and 67 days
  Subjects will undergo the measurement of gingival bleeding index according to J. Ainamo.
  Data will be collected based on clinical conditions corresponding to the score related to percentage of bleeding sites:
  Score 0-1 = 0 %-100 % (bleeding)
  Change = (Score after 67 days - Baseline score)
Effect of cannabidiol on periodontal health (modified gingival index) of patients with chronic periodontitis | Baseline (0 day) and 67 days
  Subjects will undergo the measurement of modified gingival index according to R.R. Lobene.
  Data will be collected based on clinical conditions corresponding to the scoring:
  Score 0.1-1 (mild inflammation) Score 1.1-2 (moderate inflammation) Score 2.1-3 (severe inflammation)
  Change = (Score after 67 days - Baseline score)

SECONDARY OUTCOMES:
Effect of cannabidiol on oral microbiota | Baseline (0 day) and 67 days
  Evaluation of cannabidiol effect on the composition of periopathogenic bacteria (Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia (Bacteroides forsythus), Treponema denticola, Parvimonas micra, Prevotella intermedia, Fusobacterium nucleatum, Campylobacter rectus, Eubacterium nodatum, Eikenella corrodens, Capnocytophaga sp.) in oral cavity using 16s rRNA sequencing protocol. Semi-quantitative evaluation of bacterial count:
  Code (-) = no bacteria Code (+) = mild infection Code (++) = moderate infection Code (+++) = severe infection
  Change = (count after 67 days - Baseline count)
Cannabidiol oral cavity side effects and gingival immune system | Baseline (0 day) and 37 days
  Evaluation of side effects of cannabidiol based on physical examination (photodocumentation) of oral cavity and histopathological analysis of gingiva (interdental papilla), count of plasmocytes, T-lymphocytes, B-lymphocytes and macrophages) will also be performed. Finally, the inflammatory grade according to the number of inflammatory cells per field of view will be evaluated. The intensity of inflammatory response will be classified as:
  minimal inflammation (number of immune cells up to 60 per field of view), mild inflammation (number of analyzed immune cells in the range of 61 to 100), moderate inflammation (focally confluent sheets of inflammatory cells in the range of 101 to 200), severe inflammation (confluent sheets of inflammatory cells in number more than 200).
  Change = (count after 37 days - Baseline count)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dentistry, Olomouc University Hospital, Olomouc, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stahl V, Vasudevan K. Comparison of Efficacy of Cannabinoids versus Commercial Oral Care Products in Reducing Bacterial Content from Dental Plaque: A Preliminary Observation. Cureus. 2020 Jan 29;12(1):e6809. doi: 10.7759/cureus.6809. PMID 32038896
- [Background] Vasudevan K, Stahl V. Cannabinoids infused mouthwash products are as effective as chlorhexidine on inhibition of total-culturable bacterial content in dental plaque samples. J Cannabis Res. 2020 Jun 23;2(1):20. doi: 10.1186/s42238-020-00027-z. PMID 33526124
- [Background] Lowe H, Toyang N, Steele B, Bryant J, Ngwa W, Nedamat K. The Current and Potential Application of Medicinal Cannabis Products in Dentistry. Dent J (Basel). 2021 Sep 10;9(9):106. doi: 10.3390/dj9090106. PMID 34562980
- [Background] RUSSELL AL. A system of classification and scoring for prevalence surveys of periodontal disease. J Dent Res. 1956 Jun;35(3):350-9. doi: 10.1177/00220345560350030401. No abstract available. PMID 13332137
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] Ainamo J, Bay I. Problems and proposals for recording gingivitis and plaque. Int Dent J. 1975 Dec;25(4):229-35. PMID 1058834
- [Background] Lobene RR, Weatherford T, Ross NM, Lamm RA, Menaker L. A modified gingival index for use in clinical trials. Clin Prev Dent. 1986 Jan-Feb;8(1):3-6. No abstract available. PMID 3485495
- [Background] Jirasek P, Jusku A, Simanek V, Frankova J, Storch J, Vacek J. Cannabidiol and periodontal inflammatory disease: A critical assessment. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2022 May;166(2):155-160. doi: 10.5507/bp.2022.012. Epub 2022 Mar 21. PMID 35332345